CLINICAL TRIAL: NCT06096454
Title: Effect of Life Style Modification and Metformin on Hypothyroidism With Insulin Resistance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Hasan AbdEllah, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: life style in hypothyroidism
Record Dates: First submitted 2023-09-29; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hypothyroidism; Insulin Resistance
MeSH Terms: conditions — Hypothyroidism; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin ,life style (Experimental): known to have hypothyroidism with insulin resistance received metformin (1000mg,once daily per oral ) and applied life style modification
  Interventions: Drug: Metformin
- placebo (No Intervention): known to have hypothyroidism with insulin resistance not received metformin and not applied life style modification

INTERVENTIONS:
Drug: Metformin — effect of life style modification and metformin on hypothyroidism with insulin resistance
  Other Names: life style modification
  Arms: metformin ,life style

SUMMARY:
The aim of the study is the effect of lifestyle modification and metformin on hypothyroidism with insulin resistance

DETAILED DESCRIPTION:
Hypothyroidism happens when the thyroid does not create and release enough thyroid hormone in the body this make the metabolism slow down .

Thyroid hormones T3 and T4 maintain a fine balance of glucose homeostasis by acting as insulin agonistic and antagonistic. Hypothyroidism can break this equilibrium and alter glucose metabolism, which can lead to insulin resistance.

Insulin resistance is defined clinically as the inability of a known quantity of exogenous or endogenous insulin to increase glucose uptake and utilization in an individual as much as it does in a normal population.

In this work we assess the lifestyle modification (i.e. diet and exercise)and metformin on insulin resistance

ELIGIBILITY:
Inclusion Criteria:

* 1_ above 18 years with insulin resistance criteria according (The American Association of Clinical Endocrinologists (AACE)

  * 1)BMI of 25 kg/m2 or higher
  * 2)Waist circumference of more than 102 cm in men or more than 88 cm in women
  * 3)Triglyceride level of 150 mg/dl . or higher.
  * 4) HDL-C level of less than 40 mg/dl in men or less than 50 mg/dl in women
  * 5)Blood pressure of 130 /85 mmhg or higher
  * 6)Fasting glucose level of 110 ـ126 mg /dl
  * 7)Glucose level of more than 140 mg/dl2 hour after administration of 75 g of glucose

    2_ Patients known to have hypothyroidism and achieving diagnostic criteria of insulin resistance

Exclusion Criteria:

* Patients don't have other secondary causes of insulin resistance i.e. acromegaly, Cushing syndrome 3- patient have renal or hepatic impairment (contraindication to metformin )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
change of waist circumference | 6 months
  change of waist circumference from baseline and at the end of study
Dose of levothyroxine | 6 months
  change of the dose of levothyroxine
change of parameter of metabolic syndrome | 6 months
  change of score of parameter of metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad HM AbdEllah-Alawi, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts CK, Hevener AL, Barnard RJ. Metabolic syndrome and insulin resistance: underlying causes and modification by exercise training. Compr Physiol. 2013 Jan;3(1):1-58. doi: 10.1002/cphy.c110062. PMID 23720280
- [Background] Crandall JP, Knowler WC, Kahn SE, Marrero D, Florez JC, Bray GA, Haffner SM, Hoskin M, Nathan DM; Diabetes Prevention Program Research Group. The prevention of type 2 diabetes. Nat Clin Pract Endocrinol Metab. 2008 Jul;4(7):382-93. doi: 10.1038/ncpendmet0843. Epub 2008 May 20. PMID 18493227